CLINICAL TRIAL: NCT04734509
Title: Comparison of the Silhouette and Porter Brown Systems Used in Inhalation Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Haya Alzaabi, Dr, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 233026
Record Dates: First submitted 2020-12-10; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Nitrous Oxide Inhalation Sedation
Keywords: Nitrous oxide Inhalation Sedation; Silhouette Breathing System; Porter Brown Breathing system; Scavenging system; Comparison between two breathing systems; Silhouette Mask; Porter Brown Mask; Dental anxiety; Pediatric dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Porter Brown Breathing system (Experimental): The Porter Brown has a double mask system that is characterized by a mask-within-a-mask scavenging system. The system includes easy to remove inner masks which vent into the outer mask. This helps in cleaning and sterilization. The soft inner part of the mask system provides a comfortable fit and an excellent seal around the patient's nose.
  This mask is routinely used in inhalation sedation for children's dental treatment.
  This is a sterilisable system.
  Interventions: Device: Silhouette breathing system
- Silhouette Breathing system (Experimental): The Silhouette is a single-use nasal mask and breathing circuit with lightweight tubing and an adhesive strip across the bridge of the nose to secure the mask in place and create a good seal around the patient's nose.
  Interventions: Device: Silhouette breathing system

INTERVENTIONS:
Device: Silhouette breathing system — The Silhouette is a single-use nasal mask and breathing circuit with lightweight tubing and an adhesive strip across the bridge of the nose to secure the mask in place and create a good seal around the patient's nose.
  Other Names: Silhouette Mask

SUMMARY:
This is a randomised non-blinded controlled clinical trial, which involves the measurement of efficiency and acceptability of the Silhouette Mask system and compares it with the Porter Brown Mask system used for Inhalation Sedation in children having dental treatment at the Leeds Dental Institute.

All eligible participants will be introduced to both masks (Porter Brown and Silhouette) in the assessment session prior to their first treatment session. Then participants will be randomly allocated to undergo treatment under nitrous oxide-oxygen inhalation sedation using either the Porter Brown or the Silhouette System. The efficiency and acceptability will be measured by a feedback questionnaire at the end of the treatment session and the scavenging efficiency will be measured by a diffusion pen which will measure the levels of nitrous oxide in the dentist's environment

DETAILED DESCRIPTION:
This study is a "randomised non-blinded controlled clinical trial", where a total of fifty-four patients (n=54) will be recruited from the Sedation Unit (SU) at Leeds Dental Institute on the assessment appointment (1st visit). Participants will be randomly assigned to two different inhalation sedation breathing masks either the Porter Brown system or the Silhouette system on the day of the treatment session (2nd visit) using Block Randomisation. It is planned to recruit 4-6 patients every week until 54 participants are reached. On the assessment day (1st visit), Information Sheets and the procedures will be explained in details to parents and children in simplified language and questions will be answered. All participants will be introduced to both masks the Porter Brown system and Silhouette system. Then each participant will be given an appointment for the 2nd visit. On the treatment day (2nd visit), informed consent/assent will be explained and signed by those who meet the eligibility criteria. During the treatment session, a monitoring sheet will be used and data will be collected.

Prior to the start of the study a meeting will be convened with the trained sedation assistant and the lead researcher (HA) to explain the study and to introduce the breathing systems. The potential participants will be from the waiting list where patients are waiting for sedation appointments. The lead researcher who is part of the clinical care team will identify and contact those patients by sending them Information Sheets about the study through the post besides the first assessment appointment at least two weeks before the first visit.

On the assessment day (1st routine visit), Information Sheets and the procedures will be explained in details to parents and children in simple language and questions will be answered. Participants will be introduced to both masks then appointments for the 2nd visit will be given for commencement of dental treatment under inhalation sedation for patients who agreed to participate in this study. However, for the patients who did not meet the eligibility criteria or did not want to participate in the study, they will be given regular appointments for their treatment.

On the day of the treatment ( 2nd routine Visit) informed consent and assent forms will be explained and signed by those who met the eligibility criteria. Each participant will be treated under Inhalation Sedation using one of two routinely used breathing systems depending on the Block Randomization results. he participant will be asked to complete a feedback questionnaire related to the mask used which will add about 10 to 15 mins to their routine visit. Demographic Data such as Age, Gender and the treatment carried out, the Monitoring Data, Behaviour score will be collected from the patient's dental notes.

At the second visit, each participant will be treated under Inhalation Sedation using either the Silhouette or the Porter Brown mask system depending on the session Block Randomization results. Before starting the treatment session, each participant will be examined for eligibility, If the participant has a blocked nose for example, due to a common cold, he/ she will be rescheduled for another visit or otherwise the participant will proceed to have his/ her treatment session. During the treatment session, the lead researcher (HA) will setup and assemble the breathing system parts and choose the correct size of the mask for the patient. The lead researcher will also record airflow (including volume, patient breathing rate, and level of sedation) and collect participants' data.

In addition to that, the dental nurse sedation assistant will monitor the participant and record the information on the monitoring sheet. After the treatment session, the participant will be asked to complete a feedback questionnaire related to the mask used.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the sedation unit for dental treatment under inhalation sedation.
* Children aged 7 to 15 years.
* American Society of Anaesthesiologists classification (ASA) Class I or II.
* Participants who can breathe through their nose/ no upper respiratory tract problems including large adenoids/tonsils.
* Able to follow and comply with instructions.
* First time using inhalation sedation.

Exclusion Criteria:

* Participants who are not able to communicate directly with the health care personnel carrying out the treatment.
* Uncooperative participants who refuse treatment on the dental chair.
* Participants who can't breathe through their nose (Mouth breathers).
* Participants who refuse to wear the mask.
* American Society of Anaesthesiologists classification ASA III and IV

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
The scavenging efficiency of the two breathing systems | through study completion, Up to an average of 1 year
  Its will be measured by calculating nitrous oxide levels in the ambient air using diffusion tubes. Diffusion tubes/pens work by molecular diffusion. The compound in the air has higher concentration than the tube, therefore compounds diffuse into the tube and collect on the absorbent at the end of the tube.
  At the end of the sampling period, the pens will sealed by the lead researcher (HA) and sent to Gradko Environmental Laboratory for analysis.

SECONDARY OUTCOMES:
Comfort of wearing the masks | through study completion, an average of 1 year
  Feedback about the comfort of wearing the masks (Porter Brown/ Silhouette) will be obtained from the study participants after the treatment session using a questionnaire, being developed and piloted prior to the start of the study Every child give their feedback at the end of their treatment session though a simple questionnaire
Level of patient cooperation | through study completion, an average of 1 year
  The lead researcher (HA) who will provide treatment for all participants, will assess the level of patient cooperation and record it on a data-monitoring sheet at the end of the treatment session.
  at the end of the treatment session, every child will be scored by the dentist (chief investigator)
Child dental anxiety level before and after treatment session | through study completion, an average of 1 year
  The lead researcher will assess the dental anxiety level twice before and after the treatment session and then will record it in the data-monitoring sheet.
  Dental anxiety level in children will be measured using the Facial Image Scale (FIS). This is measured twice for every child (participant), once prior the treatment started and the other one at the end of the treatment session
Mask and circuit costs of the Porter Brown and the Silhouette systems | through study completion, an average of 1 year
  The Porter Brown is a reusable system that is being sterilised between use. the cost of each breathing system will be calculated at the end of the study, and compare between the two breathing systems However, the Silhouette is a disposable system. This study will calculate the costs and compare between the two systems.

CONTACTS AND LOCATIONS:
Overall Officials: Haya Alzaabi, Prof Doc Paed Dentistry, Principal Investigator — University of Leeds, Leeds Dental Institute
Locations (1):
- Leeds Dental Institute - LTHT, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Children participants were informed that in case the study was published, their information and data will be anonymised and will not be identified.